CLINICAL TRIAL: NCT02348879
Title: A Placebo Controlled, Randomized, Double-blind, Sequential, Rising, Single Dose Study to Examine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous and Subcutaneous AMG 403 in Healthy Young and Older Adult Subjects
Brief Title: A Study to Examine the Safety, Pharmacokinetics and Pharmacodynamics of AMG 403 in Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20040195
Record Dates: First submitted 2014-12-23; First posted 2015-01-28 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — AMG 403

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 403 (Experimental): AMG 403 administered as subcutaneous and intravenous doses
  Interventions: Drug: AMG 403
- Placebo (Placebo Comparator): No active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 403 — AMG 403 is for treatment of subjects with chronic pain
  Arms: AMG 403
Drug: Placebo — contains no active drug
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety of AMG 403 in healthy adult subjects. The study consists of a 21 day screening period followed by administration of the investigational product and up to 154 day evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of non-child bearing potential,
* Between the ages of 18 and 55 inclusive,
* Body mass index from 18 to 33 kg/m2,
* Skin type compatible with the study assessments, and without significant skin allergies, pigmentary disorders, tattoos, or any active dermatologic conditions that might interfere with the study conduct.

Exclusion Criteria:

* Prior or current history of peripheral neuropathy, paraesthesias, dysesthesias, herpes zoster, post-herpetic neuralgia,
* Evidence of any current illness such as a common cold, viral syndrome, or flu-like symptoms, any disturbance of the autonomic nervous system,
* History of Raynaud's phenomenon; Know allergy or intolerance to capsaicin or hot peppers.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | up to 112 days
Incidence of abnormal clinically significant vital signs | up to 112 days
  Vital signs to be assessed included temperature, respiratory rate, pulse rate and rhythm (regular/irregular), and blood pressure. Generally, abnormal vital signs were only reported as adverse events if they required treatment or were associated with an adverse event.
Incidence of abnormal clinically significant chemistry, hematology and urinalysis test results | up to 112 days
  Laboratory abnormalities were defined by laboratory normal ranges and were not reported as adverse events unless symptomatic or associated with an adverse event.
Incidence of abnormal clinically significant ECG results | up to 112 days
  ECG abnormalities were reported as adverse events if they represented a change from baseline or if associated with symptoms or an adverse event.

SECONDARY OUTCOMES:
Pharmacokinetics profile of AMG 403 including Tmax, AUClast and Cmax | up to 112 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Gow JM, Tsuji WH, Williams GJ, Mytych D, Sciberras D, Searle SL, Mant T, Gibbs JP. Safety, tolerability, pharmacokinetics, and efficacy of AMG 403, a human anti-nerve growth factor monoclonal antibody, in two phase I studies with healthy volunteers and knee osteoarthritis subjects. Arthritis Res Ther. 2015 Oct 8;17:282. doi: 10.1186/s13075-015-0797-9. PMID 26449617
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com